CLINICAL TRIAL: NCT00602420
Title: Prevention of Pegfilgrastim-Induced Bone Pain (PIBP): A Phase III Double-Blind Placebo-Controlled Clinical Trial
Brief Title: Prevention of Pegfilgrastim-Induced Bone Pain (PIBP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Morrow, Director, URCC / University of Rochester NCORP Research Base, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CDR0000584341; U10CA037420 (NIH); URCC-07079 (Other: URCC)
Record Dates: First submitted 2008-01-22; First posted 2008-01-28 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-10

CONDITIONS: Musculoskeletal Complications; Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: pain; musculoskeletal complications; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Pain | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naproxen (Experimental): Patients receive oral naproxen twice daily beginning on the day pegfilgrastim is administered (day 2, 3, or 4) and continuing for 5-8 days.
  Interventions: Drug: naproxen
- Placebo (Placebo Comparator): Patients receive an oral placebo twice daily beginning on the day pegfilgrastim is administered (day 2, 3, or 4) and continuing for 5-8 days.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: naproxen — Oral naproxen twice daily for 5-8 days.
  Arms: Naproxen
Other: placebo — Oral placebo twice daily for 5-8 days.
  Arms: Placebo

SUMMARY:
RATIONALE: Naproxen may help prevent or lessen bone pain caused by pegfilgrastim. It is not yet known whether naproxen is more effective than a placebo in preventing bone pain caused by pegfilgrastim in patients with non-hematologic cancer undergoing chemotherapy.

PURPOSE: This randomized phase III trial is studying naproxen to see how well it works compared with a placebo in preventing bone pain caused by pegfilgrastim in patients with non-hematologic cancer undergoing chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the efficacy of daily administration of naproxen vs placebo in preventing or reducing the severity and duration of pegfilgrastim-induced bone pain (PIBP) in patients with non-hematologic malignancies undergoing chemotherapy.

Secondary

* To identify potential risk factors for the development of PIBP.
* To identify potential clinical predictors for the response or failure to respond to naproxen in preventing PIBP.
* To assess the toxicity of naproxen when administered in the preventive setting.

OUTLINE: This is a multicenter study. Patients are stratified by Clinical Community Oncology Program (CCOP) site. Patients are randomized to 1 treatment arm vs placebo.

* Arm I: Patients receive oral naproxen twice daily beginning on the day pegfilgrastim is administered (day 2, 3, or 4) and continuing for 5-8 days.
* Arm II: Patients receive matching placebo twice daily beginning on the day pegfilgrastim is administered (day 2, 3, or 4) and continuing for 5-8 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a non-hematologic (non-myeloid) malignancy
* Scheduled to receive chemotherapy; chemotherapy may be given for adjuvant, neoadjuvant, curative, or palliative intent
* Scheduled to receive the first dose of pegfilgrastim (Neulasta®) to ameliorate chemotherapy-induced neutropenia
* Creatinine ≤ 1.5 times upper limit of normal
* Able to understand English
* More than 6 months since prior surgery on the heart

Exclusion Criteria:

* Pregnant or nursing
* Clinical evidence of active gastrointestinal bleeding, prior gastrointestinal bleeding, or gastric or duodenal ulcers
* Allergy to naproxen
* Prior development of the triad of asthma, rhinitis, and nasal polyps after taking acetylsalicylic acid (aspirin) or other NSAIDs
* Concurrent nonsteroidal anti-inflammatory drugs (NSAIDs), such as aspirin, ibuprofen, or any product containing naproxen (e.g., Naprosyn, EC-Naprosyn, Anaprox, Anaprox-DS, Naprosyn suspension, or Aleve), on a regular basis
* Concurrent steroids on a regular basis
* Concurrent prescription or non-prescription medications for preexisting chronic pain; concurrent cardioprotective doses (≤ 325 mg/day) of aspirin allowed
* Concurrent therapeutic doses of warfarin

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2008-06; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Kirshner, MD, Study Chair — CCOP - Hematology-Oncology Associates of Central New York; Gary R. Morrow, PhD, MS, Study Chair — University of Rochester; Jeffrey K. Giguere, MD, FACP, Study Chair — CCOP - Greenville
Locations (16):
- United States (16):
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naproxen | Placebo
Started | 257 | 253
Completed | 232 | 229
Not Completed | 25 | 24
Not completed — Death | 1 | 4
Not completed — Chemotoxicity, Inc. Data,Ineligible | 5 | 3
Not completed — Withdrawal by Subject | 18 | 17
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: At least 145 evaluable patients in each treatment group, thus 290 evaluable patients in total, required for an 80% power analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen | Placebo | Total
Number analyzed (Participants) | 257 | 253 | 510
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (12.8) | 56.8 (11.1) | 56.2 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants] — 86% female, 14% male patients.
  Participants
    Female | 222 | 215 | 437
    Male | 35 | 38 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 19 | 33
  White | 228 | 227 | 455
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 257 | 253 | 510
Tumor Type [Number; unit: participants] — Patients required to have diagnosis of nonmyeloid cancer and were approached for study participation before first dose of pegfilgrastim on day 2, 3, or 4 of chemotherapy cycle.
  participants
    Breast | 175 | 166 | 341
    Gynecologic | 16 | 13 | 29
    Hematologic | 18 | 17 | 35
    Lung | 22 | 31 | 53
    Other | 26 | 26 | 52
Marital Status [Number; unit: participants]
  Married | 181 | 179 | 360
  Not Married | 72 | 72 | 144
  Unknown | 4 | 2 | 6
Education [Number; unit: participants]
  Some college | 180 | 164 | 344
  High school or less | 73 | 87 | 160
  Other | 4 | 2 | 6
Previous tamoxifen [Number; unit: participants]
  Yes | 8 | 11 | 19
  No | 245 | 240 | 485
  Unknown | 4 | 2 | 6
Previous chemotherapy [Number; unit: participants]
  Yes | 60 | 75 | 135
  No | 193 | 176 | 369
  Unknown | 4 | 2 | 6
Previous Radiation Therapy [Number; unit: participants]
  Yes | 18 | 30 | 48
  No | 235 | 221 | 456
  Unknown | 4 | 2 | 6
Pain at its worst in last 24 hours (scale, 0-10) [Mean (Standard Deviation); unit: units on a scale] — Any rating of bone pain from 1 to 10 was considered a day with pain. "No pain" is an instance in which patients scored their pain 0, and "any pain" for all other responses. Severe pain was similarly defined as any bone pain score greater than 5.
  units on a scale | 1.78 (2.24) | 1.87 (2.23) | 1.83 (2.24)
Bone pain today or during previous 3 days (scale, 0-10) [Mean (Standard Deviation); unit: units on a scale] — Any rating of bone pain from 1 to 10 was considered a day with pain. "No pain" is an instance in which patients scored their pain 0, and "any pain" for all other responses. Severe pain was similarly defined as any bone pain score greater than 5.
  units on a scale | 0.47 (1.44) | 0.64 (1.60) | 0.56 (1.52)

OUTCOME MEASURES:

1. Primary Outcome: Area Under Curve (AUC) of Average Pain From Diary vs. Day (1-5), Calculated by the Trapezoidal Rule.
Description: Severity and duration of bone pain (day 1 being the day pegfilgrastim is administered) as measured by a daily diary. Patients recorded daily pain (Pain Scale Score) severity on a scale of 0 (no pain) to 10 (pain as bad as you can imagine) for the last 24 hours. The AUC range was 0-40, and the units are (Pain Scale Score)*Days.
Time Frame: From baseline through day 5
Measure: Mean (95% Confidence Interval); unit: (Pain Scale Score)*Days
Arm/Group | Naproxen | Placebo
Number analyzed (Participants) | 232 | 229
(Pain Scale Score)*Days | 6.04 [4.94 to 7.14] | 7.71 [6.59 to 8.84]
Statistical Analysis 1: Comparison: Naproxen vs Placebo; Tested at the two-sided 0.05 significance level; Test type: Superiority or Other; p = 0.037, t-test, 2 sided; Mean Difference (Final Values) = 1.67, 95% CI 2-sided [0.10 to 3.24]
Statistical Analysis 2: Comparison: Naproxen vs Placebo; Tested at the two-sided 0.05 significance level; Test type: Superiority or Other; p = 0.007, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Naproxen | Placebo
Serious Adverse Events (participants affected / at risk) | 5/257 | 3/253
Other Adverse Events (participants affected / at risk) | 4/257 | 3/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naproxen (N=257) | Placebo (N=253)
Death (General disorders) | 5 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen (N=257) | Placebo (N=253)
Supraventricular tachycardia (SVT); Rash (Cardiac disorders) | 1 (1) | 0 (0)
Infection - right breast w/ cellulitis, normal ANC (Infections and infestations) | 1 (1) | 0 (0)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Acute pain secondary to marrow expansion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hospitalized d/t NV, Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutropenic fever (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No